CLINICAL TRIAL: NCT05652309
Title: Obturator Block in Lateral Tumors of the Bladder: Does it Have Adverse Effects on Early Postoperative Mobilization?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Serap Diker, Anesthesiology and Reanimation, Ankara City Hospital Bilkent
Other Study IDs: E2-22-1854
Record Dates: First submitted 2022-12-06; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Obturator Nerve Block; Ultrasound Guided Nerve Block; Complications Neurological
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- spinal anesthesia: spinal block will be performed to patients after monitoring
  Interventions: Procedure: spinal block and obturator nerve block
- spinal anesthesia and obturator nerve block: spinal block will be performed to patients after monitoring, and then the patients in the ONB block group will be given the appropriate position, with a USG-assisted distal approach, 5 cc %2 prilocain into the anterior and 5cc %2 prilocain into the posterior branch of the obturator nerve.
  Interventions: Procedure: spinal block and obturator nerve block

INTERVENTIONS:
Procedure: spinal block and obturator nerve block — spinal block and obturator nerve block

SUMMARY:
Investigation of delay in postoperative mobilization due to motor block and complications related to block in patients who underwent USG-assisted obturator nerve block with distal approach

ELIGIBILITY:
Inclusion Criteria:

* age between 18-75
* ASA1, ASA2, ASA 3 physical status

Exclusion Criteria:

1. The patient's refusal
2. Active infection in the area to be blocked
3. Kidney failure
4. Liver failure
5. Heart failure
6. BMI less than 18 and a BMI greater than 40

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who will undergo transurethral resection of the bladder
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
pin prick test | postoperatively 2nd hour
  postoperatively sensation block
bromage score | postoperatively 2nd hour
  motorial block
pin prick test | postoperatively 5th hour
  postoperatively sensation block
bromage score | postoperatively 5th hour
  motorial block

CONTACTS AND LOCATIONS:
Locations (1):
- Serap Diker, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided